CLINICAL TRIAL: NCT06008288
Title: A Single-arm, Multicenter, Open-label Phase II Clinical Study Evaluating the Efficacy and Safety of JAB-21822 Monotherapy in Patients With Locally Advanced or Metastatic Pancreatic Cancer and Other Solid Tumors Harboring the KRAS p.G12C Mutation.
Brief Title: A Phase II Study Evaluating JAB-21822 Monotherapy in Adult Patients With Pancreatic Cancer and Other Solid Tumors Harboring the KRAS p.G12C Mutation.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JAB-21822-2001
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-10

CONDITIONS: KRAS P.G12C; Pancreatic Cancer; Solid Tumor
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JAB-21822 (Experimental): Monotherapy
  Interventions: Drug: JAB-21822

INTERVENTIONS:
Drug: JAB-21822 — 800mg, orally QD with 21 days each cycle, treatment till disease progression or intolerable toxicity or withdraw for other reasons
  Other Names: Glecirasib

SUMMARY:
Patients with other advanced solid tumors (excluding NSCLC and CRC) who have progressed after prior systemic therapy or are intolerant and lack satisfactory alternative treatment options, aiming to evaluate the efficacy and safety of Glecirasib in these patients.

DETAILED DESCRIPTION:
This study is a single-arm, multicenter, open-label, basket-design, pivotal phase II trial targeting adult patients with locally advanced or metastatic solid tumors harboring the KRAS p.G12C mutation. The included populations are:

* Patients with advanced pancreatic cancer who have progressed or are intolerant to prior gemcitabine-based chemotherapy regimens or FOLFIRINOX/mFOLFIRINOX/NALIRIFOX treatments.
* Patients with other advanced solid tumors (excluding NSCLC and CRC) who have progressed after prior systemic therapies or are intolerant and lack satisfactory alternative treatment options.

The study aims to evaluate the efficacy and safety of Glecirasib in these patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the KRAS p.G12C mutation confirmed through testing using prospectively validated companion diagnostic reagents or clinical trial assay (CTA) methods.
* Histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumors (excluding NSCLC and CRC).
* Patients with pancreatic cancer must have progressed or been intolerant to prior gemcitabine-based chemotherapy regimens or FOLFIRINOX/mFOLFIRINOX/NALIRIFOX treatment. Patients with other types of solid tumors must have progressed or been intolerant to prior systemic therapies and lack satisfactory alternative treatment options.

Exclusion Criteria:

* Previously received a KRAS G12C inhibitor.
* History of interstitial lung disease, non-infectious pneumonia, or uncontrolled lung disease (including pulmonary fibrosis, acute lung disease, etc.) with clinical symptoms.
* Uncontrolled pleural effusion, pericardial effusion, or ascites.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 electrocardiograms.
* Use of a drug with known risk of torsades de points (TdP) within 14 days prior to the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by independent central radiological review (IRC) according to RECIST 1.1. | Approximately 1.5 years
  ORR is defined as the proportion of participants with confirmed complete response or partial response by IRC according to RECIST 1.1.

SECONDARY OUTCOMES:
Duration of response (DOR) | Approximately 1.5 years
  DOR is defined as the time from date of the first objective tumor response (CR or PR) to the first documentation of either Progression of Disease (PD) or death due to any cause, whichever occurs first.
Time to response (TTR) by IRC according to RECIST 1.1 | Approximately 1.5 years
  TTR is defined as the duration of time between the date of the first dose and the date of first documented response of either CR or PR.
Progression-free survival (PFS) by IRC according to RECIST 1.1 | Approximately 1.5 years
  PFS is defined as time from the first dose until disease progression or death from any cause, whichever occurs first.
Disease control rate (DCR) by IRC according to RECIST 1.1 | Approximately 1.5 years
  DCR is defined as the proportion of participants with BOR of CR or PR or stable disease (SD)
CA19-9 response rate (Applicable only to pancreatic cancer) | Approximately 1.5 years
  CA19-9 response rate is defined as the proportion of participants with CA19-9 response (achieving ≥50% decrease in CA19-9 serum levels).
Overall survival (OS) | Approximately 2.0 years
  OS is defined as time from date of the first dose to date of death due to any cause.
Number of participants with adverse events | Approximately 1.5 years
  Participants will be assessed for incidence and severity of AEs according to NCI-CTCAE 5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Shanghai Allist Pharmaceuticals, Study Director — Shanghai Allist Pharmaceuticals Co.,Ltd.
Locations (31):
- China (31):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun, Yat-sen University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute＆Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang